CLINICAL TRIAL: NCT05112458
Title: Pilot Randomized Control Trial of Cope 360 App for Caregivers of Children With Cancer
Brief Title: Cope 360 App for Caregivers of Children With Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant funding ended prior to enrolling any participants.
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Emily L Mueller, Principle Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11097; 5K08CA230218-04 (NIH)
Record Dates: First submitted 2021-09-08; First posted 2021-11-08 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Cancer
Keywords: mobile health; supportive care; adolescent; child; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Half of the participants will receive the intervention and half will receive standard care. All will be assessed at enrollment, 1 month, 3 month, and 6 month time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cope 360 application (Experimental): Participants are given access to the application and will use it to care for their child with cancer for a period of 6 months.
  Interventions: Other: Cope 360 mobile health application
- Usual Care (Active Comparator): Participants are given usual care and not given access to the application. They will be surveyed along with the experimental group for a period of 6 months.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Cope 360 mobile health application — Cope 360 is a mHealth (mobile health) app designed to support caregivers of children with cancer with symptom tracking, medication management, and emergency preparedness. We will evaluate Cope 360 via a pilot, randomized control trial in which some caregivers will receive the app and some will not. The purpose of this study is to assess: 1) feasibility of caregiver use over extended period of time, 2) acceptability of the mHealth tool by caregivers in a real-world setting, 3) impact of the mHealth tool on caregiver self-efficacy, mastery of caregiving skills/knowledge, and caregiver stress, and 4) effect on healthcare utilization of the child with cancer (i.e. preliminary data about sick visits and ED encounters).
  Arms: Cope 360 application
Other: Usual care — Caregivers of children with cancer will receive the usual clinical care provided to our patient population.
  Arms: Usual Care

SUMMARY:
To date, most caregiver focused interventions have been targeted at caregivers of adults with cancer, completely ignoring the unique needs of caregivers of children with cancer. A recent meta-analysis indicated that although these interventions had small to medium effects, they significantly reduced burden, improved ability to cope, increased self-efficacy, and improved aspects of caregivers' quality of life. Yet, several recent reviews highlighted a lack of interventions to provide practical skills for the day-to-day provision of care. The investigators have developed a pediatric oncology caregiver-focused intervention that seeks to improve caregiver clinical skills/knowledge, self-efficacy, and support seeking skills.

Cope 360 is a mHealth (mobile health) app designed to support caregivers of children with cancer with symptom tracking, medication management, and emergency preparedness. The investigators propose to evaluate Cope 360 via a pilot, randomized control trial in which some caregivers will receive the app and some will not. The purpose of this study is to assess: 1) feasibility of caregiver use over extended period of time, 2) acceptability of the mHealth tool by caregivers in a real-world setting, 3) impact of the mHealth tool on caregiver self-efficacy, mastery of caregiving skills/knowledge, and caregiver stress, and 4) effect on healthcare utilization of the child with cancer (i.e. preliminary data about sick visits and ED encounters).

DETAILED DESCRIPTION:
Procedure: The investigators will identify approximately 164 primary caregivers of children with cancer, 82 for both the intervention group and the usual care group. Those in the intervention group will be presented with the mHealth app and with the help of the RA, the participants will download the app onto their personal smartphone. Participants will be asked to use the app for a 6-month period of time. They will also receive standardized education that is provided to all caregivers of newly diagnosed patients at the investigator's institution. Those in the usual care group will receive standardized education. These caregivers will NOT be provided with access to the app.

After a participant has been enrolled in the study, the RA will collect demographic and contact information and will administer baseline assessments. Follow-up surveys with a unique identifier will be administered via email at 1, 3 and 6 months for caregivers in both the intervention and control groups. If a survey is not completed, the RA will attempt to contact the participant by phone. Surveys will be administered via Qualtrics. The investigators will collect data via these surveys on participant demographics and mobile technology usage, and outcomes will be measured utilizing the following assessments: the Caregiver Self-Efficacy scale, Caregiver Mastery scale, Pediatric Inventory for Parents, and the Technology Acceptance Model. Semi-structured interviews will be done with a subset of participants in the intervention group at the 6-month mark. Intervention participants will be contacted by phone or email and asked to participate in the interview until a subset of 30 is reached. Interviews will be conducted in person, by phone, or by Zoom videoconferencing depending on the clinic schedule of the participant's child.

Randomization: Caregivers will be randomized into either the intervention group or the usual care group. Randomization tables will be generated with SAS v9.4 utilizing the PROC PLAN procedure.

Data Collection and Analysis: Data will be collected on a variety of socio-demographic factors that have been hypothesized to impact acceptability and use of technology: age, education, gender, race, income, prior experience/exposure/awareness with computer or health technology. Information gathered will also include basic information about their child's cancer diagnosis including: type of cancer, date of diagnosis, and type of treatment protocol. Semi-structured interviews will transcribed and analyzed using Nvivo qualitative research software. Survey data will be analyzed with SAS v9.4, Qualtrics, and Microsoft Excel.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking (app is in English)
* Caregiver (parent, legal guardian, grandparent, etc.) to a child with cancer
* Caregiver to a child with cancer currently undergoing therapy (chemotherapy, radiation, etc.)
* Caregiver to a child with cancer who anticipates therapy to continue for 6 months after recruitment
* Caregiver to a child with cancer between the ages of 0 and 21 years old
* Must own a smartphone or other internet capable mobile device

Exclusion Criteria:

* Non-English speaking (app is in English)
* Caregiver with a child with cancer who is not currently undergoing therapy
* Caregiver to a child with cancer who does not anticipate therapy to continue for 6 months after recruitment
* Caregiver with a child over age 21
* Caregiver who do not own a smartphone or other internet capable mobile device

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Technology Feasibility Scale Rating | 6 months
  Feasibility of participant use over an extended period of time; measured using the Technology Acceptance Model (TAM).
Qualitative Technology Feasibility | 6 months
  Feasibility of participant use over an extended period of time; measured using semi-structured qualitative interviews.
Data Log User Acceptability | 6 months
  Acceptability by caregivers in a real-world setting; measured using audits of usage data and recorded or reported errors from data logs.
Self-Efficacy Scale Rating | 6 months
  Caregiver self-efficacy, measured using the Caregiver Self-Efficacy scale.
Mastery of Caregiving Scale Rating | 6 months
  Mastery of caregiving skills/knowledge; measured using the the Caregiver Mastery scale.
Stress Reduction Scale Rating | 6 months
  Reduction in caregiver stress; measured using the Pediatric Inventory for Parents assessment scale.
Healthcare Utilization Effect | 6 months
  Effect on healthcare utilization of the child with cancer (i.e. preliminary data about sick visits and ED encounters).

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Mueller, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT05112458/ICF_000.pdf